CLINICAL TRIAL: NCT04317950
Title: Cortical Activity During Sensorial Tactile Stimulation in Healthy Adults. The Innate Patron Activation With Vojta Therapy.
Brief Title: Cortical Activity During Vojta Stimulation in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josue Fernandez Carnero (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Clinical Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UEMURJC
Record Dates: First submitted 2020-02-28; First posted 2020-03-23 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Brain
Keywords: Electroencephalography; Electromyography; Tactile stimulation; Vojta therapy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta group (Other): All participants were properly instructed and signed an informed consent previous to the interventions. They were comfortably laid down on their back with eyes open, wearing the EEG cap and electromyography electrodes during the intervention. They were asked to remain relaxed and still during the whole process. After a first minute of resting, the experimental group received a continuous reflex locomotion stimulus during the next 8 minutes.
  Interventions: Other: Vojta
- Control group (Sham Comparator): On the contrary, the control group received a continuous sham stimulus during the next 8 minutes.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Vojta — Reflex locomotion stimulus
  Arms: Vojta group
Other: Sham — sham stimulus
  Arms: Control group

SUMMARY:
The present study is focused on the importance of sensory stimuli at the tactile and proprioceptive level that occur during the activation of the pectoral area, following the treatment protocol of Vojta Therapy (VT), and which are the areas that are activated in the central nervous system (CNS) during stimulation, as well as muscle activity. For the activation record it will be used electroencephalography and electromyography electrods.

DETAILED DESCRIPTION:
The relationship between intrinsic and extrinsic factors condition the development of the human being. The sensory organs are the main recipients of the information, thanks to them we are able to interact with the environment and register the influence of the stimuli inside the organism. The brain receives information from the environment through its senses.

At the tactile level the brain receives afferent information thanks to the activation of mechanoreceptors of the skin during interaction with the environment. The receivers encode the stimulus information and send it to the specific CNS structures. In these structures, the sensations received are combined and the stimulus is transformed into a perfectly elaborated response, both in a conscious and innate way.

Dr. Vojta showed in 1974 the locomotion reflects the result of the study of motor ontogenesis. This discovery was the demonstration of the existence of innate and preprogrammed motor patterns in Humans.

Most of the studies related to VT have showed the improvements obtained by the patients, validating it as a method of treatment and evidencing objective changes after its application. This research aim to go further and verify that cortical areas are activated during the application of an external and proprioceptive stimuli that are performed during the first phase of VT turning and which areas are responsible for producing and organizing the efferent response.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult population with no history of neurological disease or others that may affect the test.
* Age between 18 and 50 years.
* Not having addiction to alcohol or drugs at the time of the study.
* Not knowing the basics of Vojta Therapy, or knowing the responses of stimuli when applying therapy.
* Not having the pharmacological treatment that affects the functioning of the Central Nervous System and may interfere with the test results.

Exclusion Criteria:

* Those who do not meet the inclusion criteria
* Not having suffered ms-skeletal alterations in the last 6 months.
* Known sensory abnormalities.
* Diagnosis of some neurological pathology or condition that could alter the study such as pain, radiculopathy.
* Refuse to sign the informed consent.
* Claustrophobia.
* Those that can spoil the magnetic resonance image.

  * Be a carrier of some metallic material.
  * Pregnancy or nursing mother.
* The contraindications of Vojta Therapy.

  * Acute diseases that present with fever and / or inflammation.
  * Vaccination with live germs, according to medical criteria (usually 10 days after vaccination).
  * In case of crystal bone disease, uncontrolled heart disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) | 10 minutes per patient
  EEG power in alpha and beta bands
Electromyography (EMG) | 10 minutes per patient
  EMG power in Rectus abdominis, wrist extensors and tibialis anterior

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Sanz, PhD, Principal Investigator — UEM
Locations (1):
- Roberto Cano de la Cuerda, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanz-Esteban I, Cano-de-la-Cuerda R, San-Martin-Gomez A, Jimenez-Antona C, Monge-Pereira E, Estrada-Barranco C, Serrano JI. Cortical activity during sensorial tactile stimulation in healthy adults through Vojta therapy. A randomized pilot controlled trial. J Neuroeng Rehabil. 2021 Jan 21;18(1):13. doi: 10.1186/s12984-021-00824-4. PMID 33478517